CLINICAL TRIAL: NCT02891473
Title: Impact of Mézières Rehabilitative Method in Patients With Parkinson's Disease: a Randomized Controlled Trial
Brief Title: A Rehabilitative Approach in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2519/15
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Parkinson's Disease
Keywords: Posture; Pain; Muscle stretching; Mézières method; Camptocormia; Trunk control
MeSH Terms: conditions — Parkinson Disease; Pain; Camptocormia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mézières Method group (Experimental): Sessions of exercises for the recovery of midline symmetry, diaphragmatic breathing exercises, stretching of the latissimus dorsi respecting the global elongation according to the Mézières Method.
  Interventions: Other: Mézières Method
- Home based exercise program group (Active Comparator): Sessions of home based exercises performed by the patients at their domicile after a training session about the exercise program made by a physiotherapy. The exercises aimed at promoting trunk control in static and dynamic position according to the specific guidelines for Parkinson's disease and proprioceptive exercises for the recovery of balance. An illustrated exercises booklet was given to the patient.
  Interventions: Other: Home based exercise program

INTERVENTIONS:
Other: Mézières Method — 10 sessions of rehabilitative treatment according to the Mézières Method, 2 sessions per week for 5 weeks, each lasting 1 hour.
  Arms: Mézières Method group
Other: Home based exercise program — 1 single training session lasting 1 hour for the explication of the rehabilitation program that the patient has to perform independently at home followed by 2 sessions of home based exercises per week for 5 weeks, each lasting 1 hour.
  Arms: Home based exercise program group

SUMMARY:
The purpose of the study is to evaluate the effectiveness of a rehabilitative approach using breathing and relaxation techniques, and specifically the elongation of the latissimus dorsi muscle according to the Mézières Method to improve balance and posture and relief pain in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis od idiopathic Parkinson's disease (according to UK Brain Bank Criteria), Hoehn-Yahr stage ≤3 (determined during "on phase"), Mini Mental State Examination (MMSE) > or = 27, no rehabilitation treatment carried out within 3 months prior to the study, diagnosis of Parkinson's disease by at least 5 years.

Exclusion Criteria:

* Dyskinesias
* Severe fluctuations "on-off"
* Modifications of anti-Parkinsonian drug therapy during the three months prior to the start of the study)
* Sensitivity deficit of the trunk or lower extremities (physical examination)
* Vestibular disorders or paroxysmal vertigo
* Previous thoracic or abdominal surgery
* Other neurological or orthopedic conditions involving the trunk or lower extremities (musculoskeletal diseases, severe osteoarthritis, peripheral neuropathy, prosthetic surgery)
* Cardiovascular comorbidities (recent myocardial infarction, heart failure, uncontrolled hypertension, orthostatic hypotension)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of Berg Balance Scale (BBS) from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It is a widely used clinical tests to evaluate static and dynamic balance of a subject. The total score is 56 (> 45 safe walking without aids/low tendency to fall, > 35 safe walking with aids). The test lasts 15-20 minutes, and includes 14 simple tasks. The success in achieving each task is evaluated assigned a score from zero (dependent) to four (independent), and the final measure is the sum of all scores. The scale is considered the gold standard for providing useful information on the predictive estimation of the risk of falls.

SECONDARY OUTCOMES:
Change of Visual Analogue Scale (VAS) from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It is a scale for the assessment of pain and it's based on a ten point scale, where 0 means no pain and 10 the greatest pain ever both at rest and during movements.
Change of Unified Parkinson's Disease Rating Scale (UPDRS) from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It consists of six parts made up of questions about the mental state, behavior and mood, ADL, motor functions, the complications of the advanced disease, the stage of the disease identified by the Hoehen and Yahr scale and the modification in the execution of the ADL trough the scale of Schwab and England. The scale is based on a metric scale from 0 (no disability) to 147 points (severe disability).
Change of Functional Gait Assessment (FGA) from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It is a 10-items scale that measures walking balance activity and it was developed from the Dynamic Gait Index (DGI) to improve reliability and decrease the ceiling effect. Each item is scored on a 3 point-scale from 0 (severe impairment) to 3 (normal deambulation). The highest possible score is 30 (normal gait function).
Change of Clinical Evaluation of Posture from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It is the evaluation of the anterior flexion of the trunk by measuring the distance fingers-floor.
Change of Modified Parkinson Activity Scale (MPAS) from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  consists of 14 items arranged into three domains, chair transfer, gait akinesia and bed mobility. Scores range from 0 (dependent) to 4 (normal) and the total possible score is 56.
Change of SF-36 Health Survey Questionnaire from baseline to 12 weeks | Baseline, 4 weeks, 12 weeks
  It is a multi-dimensional questionnaire for the evaluation of health status. It is divided into eight sub-categories that measure physical activity, limitations due to physical health and emotional state, physical pain, the perception of general health, vitality, social activities, mental health and changes in health status and two indices that summarize the overall assessment of the subject with respect to his/her physical (ISF) and mental (ISM) health.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Study Director — Sapienza University of Rome, Policlinico Umberto I hospital
Locations (1):
- Umberto I Hospital, Rome, Italy